CLINICAL TRIAL: NCT03591575
Title: Safety and Efficacy of Early-start Deferiprone Treatment in Infants and Young Children Newly Diagnosed With Transfusion-dependent Beta Thalassemia
Brief Title: Safety and Efficacy of Early Treatment With Deferiprone in Infants and Young Children
Acronym: START
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiesi Canada Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LA55-0417
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Beta Thalassemia Major Anemia; Iron Overload
Keywords: thalassemia; iron overload; chelation; deferiprone; Ferriprox
MeSH Terms: conditions — Iron Overload; Thalassemia | interventions — Deferiprone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo solution will have the same appearance and flavor as deferiprone oral solution, and will be administered at a volume matching that required for the dose of active product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Deferiprone (Experimental): Subjects in this group will receive deferiprone oral solution at a dosage up to 75 milligrams per kilogram of body weight (mg/kg) per day, divided into 3 equal doses
  Interventions: Drug: Deferiprone oral solution
- Placebo (Placebo Comparator): Subjects in this group will receive placebo solution at a volume equal to what they would receive if they were in the active arm, divided into 3 equal doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deferiprone oral solution — Liquid formulation of deferiprone, with a concentration of 80 mg/mL
  Other Names: Ferriprox
  Arms: Deferiprone
Drug: Placebo — Liquid solution that matches deferiprone oral solution in appearance and taste
  Other Names: Placebo for deferiprone oral solution
  Arms: Placebo

SUMMARY:
This study is looking at the effects of giving early treatment of deferiprone to young children with beta thalassemia who have started receiving regular blood transfusions but have not yet reached the criteria for starting on iron chelation therapy. Half the patients in the study will receive deferiprone, and the other half will receive placebo, for up to 12 months.

DETAILED DESCRIPTION:
This study will give deferiprone to infants and young children with thalassemia who have started receiving regular blood transfusions but whose iron load is not yet at the level where chelation treatment would normally begin. The purpose is to see if doing this will postpone the build-up of iron without causing serious side effects. Half the children in the study will be given deferiprone at a dose that is lower than what is normally prescribed, and the other half will be given placebo. All patients will receive the assigned product three times a day for up to 12 months. Tests for signs of iron overload will be done monthly, and a patient whose iron load reaches the level where chelation therapy would normally begin will be immediately taken out of the study and started on standard chelation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 6 months to < 10 years
2. Confirmed diagnosis of beta-thalassemia, as determined by high performance liquid chromatography (HPLC) or DNA testing
3. Started on a red blood cell (RBC) transfusion regimen, with a minimum of 2 transfusions already completed
4. Screening level of serum ferritin (SF) greater than >200 μg/L but not more than 600 μg/L. Since SF level may be impacted by the presence of infection, it must additionally be verified that the child has had no signs of infection in the previous 7 days, including the day of screening, and that the level of C-reactive protein (CRP) is no greater than 20% higher than the normal range for the patient's age. If there are signs of infection and/or the CRP level is above this threshold, the SF level must be checked again a minimum of one week later.

Exclusion Criteria:

1. Prior use of iron chelation
2. Diagnosis of hepatitis B or C, or HIV infection
3. Evidence of abnormal liver or kidney function at screening: serum alanine transaminase (ALT) level > 5 times upper limit of normal or creatinine levels >2 times upper limit of normal
4. Disorders associated with neutropenia (absolute neutrophil count < 1.5 x 10^9/L) prior to the initiation of study medication
5. A serious, unstable illness, as judged by the investigator, during the previous 3 months before screening/baseline visit including but not limited to hepatic, renal, gastro-enterologic, respiratory, cardiovascular, endocrinologic, neurologic or immunologic disease.
6. Presence of any medical condition which in the opinion of the investigator would cause participation in the study to be unwise.

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen El Alfy, MD, Principal Investigator — Ain Shams University
Locations (4):
- Egypt (3):
  - Ain Shams University Children's Hospital, Cairo
  - Pediatric Hospital of Cairo University, Cairo
  - The Clinical Research Center, Faculty of Medicine, Cairo University, Cairo
- Cipto Mangunkusumo National Hospital, Jakarta, Indonesia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deferiprone | Placebo
Started | 32 | 32
Completed | 26 (Includes 18 subjects who received 12 months of treatment, and 8 who terminated treatment early due to having reached the threshold for starting standard chelation therapy) | 31 (Includes 11 subjects who received 12 months of treatment, and 20 who terminated treatment early due to having reached the threshold for starting standard chelation therapy)
Not Completed | 6 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferiprone | Placebo | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.03 (2.42) | 2.63 (1.70) | 2.83 (2.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 20 | 21 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 29 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 26 | 29 | 55
  Indonesia | 6 | 3 | 9
Serum ferritin (µg/L) [Mean (Standard Deviation); unit: micrograms per liter] | 513.84 (236.06) | 451.69 (196.43) | 482.76 (217.68)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients in Each Treatment Group Who Still Have a Serum Ferritin Level < 1000 Micrograms Per Liter (μg/L) at Month 12
Description: Current treatment guidelines are that standard iron chelation therapy should begin after a serum ferritin level of 1000 μg/L has been reached; thus, patients who were at this level at two consecutive visits were removed from the study so that they could start on this therapy.
Time Frame: 12 months
Population: Intent-to-Treat (ITT) population. For patients who withdrew early, imputed data were used to estimate the serum ferritin values that would likely have been seen at Month 12 had they continued.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 32 | 32
Participants | 21 | 12
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Patients who reached the serum ferritin threshold at any time point prior to Month 12 were withdrawn from the study as per protocol, so that they could begin on standard chelation therapy. For these individuals, imputed data were used to estimate the values that would likely have been seen at Month 12 had they remained in the study; Test type: Superiority; p = 0.0446, Fisher Exact

2. Secondary Outcome: Percentage of Patients With Serum Ferritin Still Below the Threshold at Different Time Points
Description: The outcome measure was the percentage of patients in each group still below the serum ferritin threshold at Months 4, 8, and 12. Without adequate chelation therapy, most patients receiving red blood cell transfusions are likely to exceed this level within a few months. However, a safety feature of the study design was that patients who reached the serum ferritin threshold were withdrawn (i.e., so that they could begin standard chelation therapy).
Time Frame: 4, 8, and 12 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  Number of patients still below threshold at Month 4 | 29 | 28
  Number of patients still below threshold at Month 8 | 22 | 20
  Number of patients still below threshold at Month 12 | 21 | 12
Statistical Analysis 1: Comparison: Deferiprone vs Placebo; Test type: Superiority; p = 0.0446, Fisher Exact — he p-value shown here is for the difference between the groups at Month 12

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Deferiprone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 5/32 | 2/32
Other Adverse Events (participants affected / at risk) | 29/32 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=32) | Placebo (N=32)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=32) | Placebo (N=32)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 20 (60) | 18 (55)
Bronchitis (Infections and infestations) | 3 (3) | 6 (7)
Gastroenteritis (Infections and infestations) | 5 (5) | 4 (5)
Nasopharyngitis (Infections and infestations) | 8 (10) | 8 (14)
Pharyngitis (Infections and infestations) | 4 (5) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (18) | 5 (8)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 9 (19) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT03591575/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03591575/SAP_001.pdf
  • Informed Consent Form (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03591575/ICF_002.pdf